CLINICAL TRIAL: NCT04293081
Title: Role of Preemptive Chlorepheniramine Maleate in Reducing Postoperative Agitation After Functional Endoscopic Sinus Surgeries (FESS)
Brief Title: Preemptive Chlorepheniramine Maleate Reducing Postoperative Agitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer Nabil Abdelrahman, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R 01/2019
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Agitated; State, Acute Reaction to Stress
Keywords: chlorpheniramine maleate, Agitation, FESS
MeSH Terms: conditions — Psychomotor Agitation; Stress Disorders, Traumatic, Acute | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chlorpheniramine maleate group (Active Comparator): A total of 45 adult patients undergoing FESS procedure for sinusitis with postoperative nasal packing. Written informed consent will be obtained from all patients before randomization. Patients will be assigned to chlorepheniramine maleate group (A)
  Interventions: Drug: Preemptive chlorepheniramine maleate intravenous injection
- placebo group (Placebo Comparator): A total of 45 adult patients undergoing FESS procedure for sinusitis with postoperative nasal packing. Written informed consent will be obtained from all patients before randomization. Patients will be assigned to placebo group (A)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Preemptive chlorepheniramine maleate intravenous injection — Participants of group A will receive only one ampoule of 45.5 mg/ 2mL chlorepheniramine maleate diluted in 8 ml isotonic saline intravenous (I.V) prior to induction of general anesthesia by 30 minutes
  Arms: chlorpheniramine maleate group
Drug: normal saline — participants in group (B) will receive 10 ml isotonic saline (placebo) by the same route as control.
  Other Names: normal isotonic saline
  Arms: placebo group

SUMMARY:
The aim of the study is to identify the role of preoperative chlorepheniramine maleate on alleviating or reducing the severity of postoperative agitation following FESS procedures.

DETAILED DESCRIPTION:
A total of 90 adult patients undergoing FESS procedure for sinusitis with postoperative nasal packing. Written informed consent will be obtained from all patients before randomization. Patients will be divided equally into two groups the first 45 patients will be assigned to chlorepheniramine maleate group (A) and the other group to placebo group (B). Group assignment, preparation and administration of drugs will be performed by a junior anesthetist who is neither involved nor interested by any means in the study. Blind grouping will be kept to all including the patients themselves, until the completion of study.

Inclusion and Exclusion Criteria The inclusion criteria of these patients include adult patients (age 18- 60 years), class I-II according to American society of anaesthesiologists (ASA) physical status subjected to FESS without septoplasty. Exclusion criteria include; patients below 18 years old or over 60 years old, patients with ASA physical status class III-IV, morbid obesity with BMI > 30 kgm-2 at initial hospital visit, history of neuro-psychatric ailment or chronic use of antipsychotic drugs, severe cardiovascular disease, any coagulopathies, pregnancy, history of relevant drug allergy, any possibility of anticipated difficult intubation.

Preoperative Anesthetic Assessment All patients will be subjected to a thorough medical history, physical examination, laboratory investigations (fasting blood sugar, kidney, liver function tests, serum electrolytes, coagulation profile, and electrocardiogram) preoperatively. They will be also counseled about the anesthetic management and potential complications of both surgery and anesthesia, and the explanations of numerical pain analogue scale (NAS) from 0-10. All these data will be documented. A thorough airway assessment by Mallampati classification, mouth opening, neck movement, thyromental distance will be done to find out any possibility of difficult intubation. If there is a chance of significant difficult intubation, the patient will be excluded from the study.

Anesthetic Protocol All patients admitted to OR induction area where patient identification is confirmed and an 18-gauge intravenous cannula will be inserted to all Participants. Participants of group A will receive only one ampoule of 45.5 mg/ 2mL chlorepheniramine maleate diluted in 8 ml isotonic saline intravenous (I.V) prior to induction of general anesthesia by 30 minutes while participants in group (B) will receive 10 ml isotonic saline (placebo) by the same route as control.

General anesthesia will be started for all patients with intravenous lignocaine 1.0 mg/kg, propofol 2.0 mg/kg, then atracurium 0.5 mg/kg, fentanyl 1 µg/kg then they will be intubated orally which is fixed after confirmation of its place by auscultation then oral packing with wet gauze under vision using laryngoscope. Anesthesia will be maintained by mixture of O2 and air along with 2% sevoflurane then atracurium 0.1 mg/kg will be given for maintenance of muscle relaxation.. All patients will be monitored by standard monitors including, the pulse oximeter, non-invasive blood pressure, end-tidal C02, and electrocardiogram. Moreover, bispectral index monitor is used to assess depth of general anesthesia.

Deliberate hypotension will be done using intravenous infusion of nitroglycerine at a rate of 5 to 20 µg/ kg /minute titrated to target mean arterial blood pressure (Mbp) of 55±5 mmHg. Hypotensive anesthesia will be maintained throughout the surgical procedure. At the end of surgery, mean arterial blood pressure (Mbp) will be elevated by stoppage of nitroglycerine infusion and infusing crystalloids (500-1000ml) together with administration of ephedrine hydrochloride 10 mg IV to restore the mean arterial blood pressure back to the preoperative value. Upon attaining spontaneous breathing muscle relaxant will be antagonized by 50 µg/kg neostigmine and 10 µg/kg glycopyrolate, then oral pack will be removed under vision with thorough oral suctioning then awake extubation will be done and the patients will be transferred to the recovery unit.

Postoperative Analgesic Regimen It will start immediately on arrival to the recovery unit where patients received 16 mg lornoxicam slowly IV over 5 minutes. After that all patients will receive acetaminophen 1 gm/6 h IV and 5 mg Nalbuphine IV if breakthrough pain develops for the first day postoperative.

Patients Assessment Patients will be transferred to Post-anesthesia care unit PACU for observation and assessment for agitation and pain. Upon arrival to PACU, a pulse oximeter and Non invasive blood pressure (NIBP) monitors will be attached to the patient. Discharge criteria from PACU will be stable vital signs, pain score less than or equal to 2, no nausea or vomiting, calm and alert patient.

Assessment of agitation Postoperative agitation will be assessed in the PACU by a blinded observer using the Richmond Agitation Sedation Scale (RASS) as follows: 0= Alert and calm +1= Restless; Anxious and /or apprehensive but movements not aggressive. +2= agitated; Frequent non-purposeful movement. +3= very agitated; Pulls on or removes the tubes or catheters or has aggressive behavior toward staff. +4= combative; overly combative or violent. Total agitation will be defined as the algebraic sum of agitation values will be observed at the measured time points (0, 5, 10, 15, 30 minutes after recovery), and this will be used to correlate agitation with other variables. The agitations score range will be from 0= no agitation to 20= severe persistent agitation.

In case of severe persistent agitation with RASS > 12 in the first 15 minutes postoperatively patients will be reassured and midazolam 2 mg IV will be given to reduce agitation with thorough follow up of patient's breathing.

Assessment of pain Pain intensity will be assessed as a secondary outcome to the investigator's study using visual analogue scale where 0= no pain and 10 is the worst imaginable pain as rated by the patient. A blinded team member assessed pain after evaluation of last agitation point (30 minutes of recovery). Patient that exhibited no agitation will be also evaluated for pain after 30 minutes of recovery. Nalbuphine will be used as rescue analgesic to ameliorate pain. The use of nalbuphine after evaluation of agitation and assessment of pain to avoid perplex to the outcome measurement. If pain is more than +6 on VAS Nalbuphine will be given in 5 mg until pain score < 4. Pain assessment is done after 2, 6 , 12 and 24 hours postoperatively with calculating the frequency of rescue analgesia given and the total dose of nalbuphine consumed during that time taking care not to exceed 5 Mg at a time with drug lag of at least 2 hours between 2 successive doses of rescue agent.

The primary end point to this study is the occurance of severe agitation endangering the patient, or the occurance hypoxemia, bleeding nasal or oral, or the occurance of postoperative atypical hypotension.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of these patients include adult patients (age 18- 60 years), class I-II according to American society of anaesthesiologists (ASA) physical status subjected to FESS without septoplasty.

Exclusion Criteria:

* Exclusion criteria include; patients below 18 years old or over 60 years old, patients with ASA physical status class III-IV, morbid obesity with BMI > 30 kgm-2 at initial hospital visit, history of neuro-psychatric ailment or chronic use of antipsychotic drugs, severe cardiovascular disease, any coagulopathies, pregnancy, history of relevant drug allergy, any possibility of anticipated difficult intubation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
reduction of postoperative agitation following FESS procedures using chlorpheniramine maleate | Start immediately postextubation (0) minute and every 5 minute for 30 minutes after recovery),
  agitation assessed by Richmond Agitation Sedation Scale (RASS)(0= alert calm, 1=restless, 2 mild agitation, 3= severe agitation, 4= combative)

SECONDARY OUTCOMES:
pain assessement: visual analogue score | starting at 30 minutes postoperative then at 2, 6, and 12 hours postoperatively
  visual analogue score( 0= no pain, 10= the worst imaginable pain)
The duration of surgery and anesthesia with time needed for extubation | intraoperative
  feasability of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams University, Faculty of medicine, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No